CLINICAL TRIAL: NCT05613647
Title: Concordance Study of Therapeutic Decision-making in Patients With Acute Circulatory Failure Between Cardiac Output Monitoring by Transthoracic Echocardiography and by Transpulmonary Thermodilution : PICC-ECHO Study
Brief Title: Concordance Study of Therapeutic Decision-making in Patients With Shock Based on Hemodynamic Monitoring
Acronym: PICC-ECHO
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022-A02017-36
Record Dates: First submitted 2022-10-30; First posted 2022-11-14 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Shock; Acute Circulatory Failure; Hemodynamic Monitoring
Keywords: hemodynamic monitoring; Concordance of decision
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Shock is a serious complication corresponding to acute circulatory failure resulting in multiorgan failure and death. In order to improve cellular oxygen utilization, several therapies can be used. To select one of them, the monitoring of cardiac output is helpful. However, there are several methods used in current practice in intensive care for evaluating hemodynamic.

Currently, in patients with acute circulatory failure, no study has compared the concordance of therapeutic decision-making based on transpulmonary thermodilution or transthoracic echocardiography.

The objective of the PICC-ECHO study is thus to assess the concordance of therapeutic decision-making by several experts, based on data from transpulmonary thermodilution or transthoracic echocardiography.

Indeed, the investigators hypothesize that performing hemodynamic monitoring based on transpulmonary thermodilution or transthoracic echocardiography does not lead to the same therapeutic management in patients in shock.

DETAILED DESCRIPTION:
PICC-ECHO is a monocentric, prospective, non interventional, exploratory study to assess the concordance of therapeutic decision-making between two strategies used in current practice, transthoracic echocardiography and transpulmonary thermodilution, in patients with acute circulatory failure.

Each patient in shock with cardiac output monitoring by transpulmonary thermodilution is identified and then eligible for inclusion.

After inclusion, measurements of cardiac output with PICCO device and transthoracic echocardiography will be performed before and after a passive leg raising test and a respiratory occlusion test if patient are under invasive mechanical ventilation.

These assessments will be conducted by two different investigators, to be sure that data by transthoracic echocardiography will not be influenced by the measurements collected by the analysis of the transpulmonary thermodilution.

Clinical, biological, echocardiographic and transpulmonary thermodilution data will be then collected on a database.

The therapeutic management of the clinicianresponsible for the patient will also be collected.

The database will be used as support for the drafting of three medical observations for each patient on an electronic CRF : one with data from transpulmonary thermodilution, one with data from transthoracic echocardiography, and one with only clinico-biological parameters (without advanced monitoring).

At the end, 45 different files will be compiled and submitted to different intensive care physicians (between 10 and 20) working outside the investigative team (" experts ").

In order to avoid any recognition between the three versions of a same patient, the investigators will undergo a semantic variation and the mailings will be done in three distinct groups corresponding to the three methods separated by a few weeks.

For each clinical case, experts will have to choose about the following choices: volume expansion, increase norepinephrine, introduction or increase dobutamine, abstention with continuation of current therapy.

Vital status of the patient as well as the use of supportive care (mechanical ventilation, renal-replacement therapy, vasoactive drug, other assistance) and their duration will be collected at day n°28.

For each case, the investigators will evaluate the concordance of decision of each expert, depending on whether the informations was collected by PICCO device, by echocardiography or without invasive monitoring.

ELIGIBILITY:
Inclusion Criteria:

* adult patient, hospitalized in the Intensive Care Medicine, CHU of Angers;
* patient requiring a hemodynamic evaluation because of an acute circulatory insufficiency defined by : arterial hypotension requiring vasopressor amines, with clinical signs (mottling, encephalopathy, oliguria > 2h) and/or biological signs (pH <7.38; lactate > 2 mmol/L) of tissue hypoperfusion;
* patient monitored by transpulmonary thermodilution with pulse wave contour measurement (PiCCO) as part of routine care.

Exclusion Criteria:

* patient with acute pulmonary heart on TTE (defined as a LV-to-VG ratio > 0.6 associated with a paradoxical interventricular septum);
* patient objecting to participation in the research;
* a relative who has received the information, if the patient's condition does not allow it, and who objects to the participation of his or her relative in the research;
* persons protected by law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient in intensive care unit for shock with cardiac output monitoring by transpulmonary thermodilution and with hemodynamic instability
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Intra-expert concordance of therapeutic management according to PICCO device or echocardiography monitoring. | at inclusion
  the concordance of hypothetical therapeutic decision-making done a posteriori by experts in patients with acute circulatory failure between cardiac output monitoring by transthoracic echocardiography or by transpulmonary thermodilution.

SECONDARY OUTCOMES:
Inter-expert concordance of therapeutic management according to PICCO device or echocardiography monitoring. | at inclusion
  the inter-expert concordance of therapeutic management according to data from transpulmonary thermodilution or transthoracic echocardiography.
Intra and inter expert concordance of therapeutic management according to PICCO device or without advance cardiac output monitoring. | at inclusion
  the intra-expert and inter-expert concordance of theoretical therapeutic management according to data provided by PICCO device or without cardiac output monitoring
History and clinical situation | at inclusion
  the difference in history and clinical situation in patients for whom theoretical therapeutic management is discordant or not according to the different methods: PICCO device vs echocardiography; PICCO vs no hemodynamic monitoring; echocardiography vs no hemodynamic monitoring
Decision of volume expansion | at inclusion
  the intra-expert and inter-expert concordance of the decision of volume expansion according to data from the different methods: PICCO vs echocardiography, PICCO vs no hemodynamic monitoring, echocardiography vs no hemodynamic monitoring
frequency of volume expansion, change in norepinephrine and dobutamine according to the method of cardiac output monitoring. | at inclusion
  the frequency of use of volume expansion, vasopressor support and inotropic support (dobutamine) according to the method of cardiac output monitoring: PICCO vs echocardiography, PICCO vs no hemodynamic monitoring, echocardiography vs no hemodynamic monitoring
the description of the expert population | at inclusion
  Description of the expert population (seniority in the intensive care unit, place of practice : hospital or university hospital, number of beds in the intensive care unit in which the expert works, which haemodynamic monitoring tool is used in current practice by the expert.
the concordance between experts and clinician management | at inclusion
  Concordance of decision between expert and clinician management

CONTACTS AND LOCATIONS:
Overall Officials: Pierre ASFAR, MD- PhD, Principal Investigator — University Hospital, Angers
Locations (1):
- CHU Angers, Angers, France